CLINICAL TRIAL: NCT00395213
Title: Antidepressant Safety in Kids (ASK) Study: An Open-label, Prospective, Cohort Study of Antidepressants in Children and Adolescents With Anxiety Disorders, Depressive Disorders, Eating Disorders, or Obsessive-Compulsive Disorder
Brief Title: Antidepressant Safety in Kids Study
Acronym: ASK
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00013655; P30MH066386 (NIH); DSIR CTM; 3159; 8067-06-1
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety Disorders; Depressive Disorders; Eating Disorders; Obsessive Compulsive Disorder
Keywords: Anxiety; Major Depression; Anorexia; Bulimia; OCD; Antidepressant; SSRI; SNRI
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Feeding and Eating Disorders; Obsessive-Compulsive Disorder; Depressive Disorder, Major; Anorexia; Bulimia | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Children and adolescents with a pre-specified anxiety disorder, depressive disorder, eating disorder, or obsessive-compulsive disorder
  Interventions: Drug: Selective serotonin reuptake inhibitor (SSRI) and serotonin-norepinephrine reuptake inhibitor (SNRI) medications

INTERVENTIONS:
Drug: Selective serotonin reuptake inhibitor (SSRI) and serotonin-norepinephrine reuptake inhibitor (SNRI) medications — Treatment with SSRIs or SNRIs

SUMMARY:
This study will evaluate the risks and benefits of treatment with a selective serotonin reuptake inhibitor or serotonin-norepinephrine reuptake inhibitor in children and adolescents with a pre-specified anxiety disorder, depressive disorder, eating disorder, or obsessive-compulsive disorder.

DETAILED DESCRIPTION:
The Antidepressant Safety in Kids (ASK) study is part of the Child and Adolescent Psychiatry Trials Network (CAPTN).

Selective serotonin reuptake inhibitor (SSRI) and serotonin-norepinephrine reuptake inhibitor (SNRI) medications are prescribed to approximately 2 to 3% of American children. Evidence suggests that these medications are beneficial for treating obsessive-compulsive disorder (OCD), anxiety disorders, and major depressive disorder. Following hearings in February and September of 2004, the FDA mandated Black Box warnings for all antidepressants, cautioning prescribers about the risk of treatment-emergent suicidal tendency in children and adolescents treated with these drugs. Although prescribing waned somewhat following the warning, many children continue to receive SSRIs and SNRIs for a variety of conditions that do not have empirically validated alternative treatments. Therefore, there is a pressing need to clearly understand the safety, tolerability, and effectiveness of SSRIs and SNRIs in children and adolescents.

Specific Aim:

The purpose of this study is to evaluate the safety, tolerability, and effectiveness of SSRI and SNRI medications for children and adolescents with anxiety disorders, depressive disorders, eating disorders, or obsessive-compulsive disorder. The study will characterize predictors of outcome, including demographic, disease severity, comorbidity, concomitant treatment, and genetic variation. This information will help clinicians to better understand the balance of risk and benefit associated with antidepressants and to answer the question of which treatment is best for which child.

Three specific aims include the following:

1. To evaluate the within-subject benefit of antidepressant treatment over acute (12 weeks) and maintenance (an additional 6 months) of treatment;
2. To evaluate the adverse event profile for harm to self, harm to others, and psychiatric and nonpsychiatric adverse events;
3. To evaluate potential moderators and mediators of benefits and adverse events.

Design:

This will be a prospective longitudinal cohort study of 2,420 consecutively enrolled patients who are prescribed an SSRI or SNRI (Citalopram [Celexa], Escitalopram [Lexapro], Fluoxetine [Prozac/Prozac Weekly], Fluvoxamine [Luvox], Paroxetine, [Paxil/Paxil-Cr], Sertraline [Zoloft], Venlafaxine [Effexor/Effexor XR], Duloxetine [Cymbalta]). Patients will be drawn from the practices of approximately 200 CAPTN participants in the United States and Canada.

Study Timeline:

This study will have two phases: 1) an acute treatment phase following initiation of treatment with any SSRI or SNRI of the clinician's choosing and 2) a long-term follow-up phase. The acute treatment phase will last 12 weeks and the long-term follow-up phase will occur 6 and 9 months after initiation of treatment.

Treatment:

Flexible upward titration of any of the commercially available SSRI or SNRI medications. As decided by the treating doctor, titration will depend on the severity of illness, degree of response, and adverse event profile. With few exceptions, concomitant treatments are permitted.

Assessment:

Study assessment milestones will occur at baseline, Week 12, and Months 6 and 9 or at study entry. CAPTN uses a "no query rule" electronic data capture system. The parent and child will complete a pen and paper workbook consisting primarily of the DISC Predictive Scales (DPS-IV) and the Pediatric Adverse Event Rating Scale (PAERS). Based on this information and on clinical interview, the treating clinician will complete the fully web-based EDC modules at baseline and at all treatment and end-of-study visits.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment in an outpatient, residential, or in-patient setting
* Meets DSM-IV diagnostic criteria for at least one of the following disorders: anxiety disorder, depressive disorder, eating disorder, or obsessive-compulsive disorder
* English- or Spanish-speaking

Exclusion Criteria:

* Inpatient status IF the enrolling inpatient clinician will not continue to follow the patient for the duration of the study
* Sibling that is already enrolled in the study
* Imminently suicidal and unable to comply with a no-suicide contract or, in the opinion of the treating clinician, has inadequate family monitoring for suicidality
* Acutely psychotic at study entry
* A demonstrated lack of benefit from or intolerance to SSRI/SNRI antidepressants, as a class
* Receiving treatment with a tricyclic antidepressant (TCA) at study enrollment, with the exception of low doses for enuresis for chronic pain. Patients may receive adjunctive TCA treatment during the study at the clinician's discretion.
* Received a monoamine oxidase inhibitor (MAOI), such as isocarboxazid (Marplan), phenelzine (Nardil), or tranylcypromine (Parnate), within the past 30 days
* Parasuicidal behavior or milder forms of suicidality or activation that do not meet the diagnostic criteria
* Refusal to participate in the pharmacogenomic study
* For bipolar depressed patients, a mixed- or manic-state at study entry without stable treatment with a mood stabilizer for manic symptoms
* Patient or family is unable to comply with the protocol

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents age 7 to 17 years old.
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Score on the Clinical Global Impression Improvement scale (CGI-I) | Measured at Months 3, 6, and 9
Clinician Patient Access to Electronic Records System | Measured at every visit
CAPTN Serious Adverse Events (SAE)/Harm-related adverse events form | Measured at every visit

SECONDARY OUTCOMES:
Score on the Clinical Global Impression Severity scale (CGI-S) | Measured at Months 3, 6, and 9
Score on the Children's Global Assessment Scale (CGAS) | Measured at Months 3, 6, and 9
Parent Coping Strategies Questionnaire (CSQ) | Measured at every visit
Youth Coping Strategies Questionnaire (CSQ) | Measured at every visit

CONTACTS AND LOCATIONS:
Overall Officials: John S. March, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Child and Adolescent Psychiatry Trials Network (CAPTN), Durham, North Carolina, United States

REFERENCES:
- [Background] March JS, Silva SG, Compton S, Anthony G, DeVeaugh-Geiss J, Califf R, Krishnan R. The Child and Adolescent Psychiatry Trials Network (CAPTN). J Am Acad Child Adolesc Psychiatry. 2004 May;43(5):515-8. doi: 10.1097/00004583-200405000-00004. PMID 15100557
- [Background] March JS, Silva SG, Compton S, Shapiro M, Califf R, Krishnan R. The case for practical clinical trials in psychiatry. Am J Psychiatry. 2005 May;162(5):836-46. doi: 10.1176/appi.ajp.162.5.836. PMID 15863782
- See also: Click here for the PARCA trial, a related study by the CAPTN network — http://www.clinicaltrials.gov/ct/show/NCT00516932